CLINICAL TRIAL: NCT07396220
Title: Combined Intranasal Esketamine and Brief Cognitive Behavioral Therapy for Suicidal Ideation - A Randomized Controlled Trial
Brief Title: Psychotherapy Combined With Intranasal Esketamine for the Treatment of Suicidal Ideation
Acronym: PIK-SI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Cory Weissman, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 813122
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Esketamine (Active Comparator): Naturalistic Intranasal Esketamine
  Interventions: Other: Naturalistic Intranasal Esketamine
- BCBT-SP + Intranasal Esketamine (Experimental): Brief Cognitive Behavioral Therapy for Suicide Prevention combined with Intranasal Esketamine
  Interventions: Other: Naturalistic Intranasal Esketamine; Behavioral: Brief Cognitive Behavioral Therapy for Suicide Prevention

INTERVENTIONS:
Other: Naturalistic Intranasal Esketamine — Naturalistic Intranasal Esketamine is administered in accordance with psychiatrist recommendations
Behavioral: Brief Cognitive Behavioral Therapy for Suicide Prevention — 12 session evidence based psychotherapy protocol with weekly 50 minute sessions
  Arms: BCBT-SP + Intranasal Esketamine

SUMMARY:
The purpose of this study is to examine the effects of combined intranasal esketamine with brief cognitive behavioral therapy for suicide prevention (BCBT-SP) for suicidal ideation (SI) in patients with treatment- resistant depression (TRD). The secondary aim is to identify the biological targets of treatment response using combined transcranial magnetic stimulation and electroencephalography (TMS-EEG). In this project we will recruit patients between the ages of 18 and 70, diagnosed with a major depressive episode with ongoing suicidal ideation present who have failed (or not shown signs of improvement) after at least one prior treatment. The null hypothesis is that there will be no difference in reductions in suicidality at 1-week post-treatment between the combined treatment group and the ketamine only treatment group. The alternative hypothesis is that the combined treatment will result in a greater reduction in suicidal ideation at 1-week post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All genders
2. Ages 18 to 70 years
3. Physician order of intranasal esketamine in the UCSD Interventional Psychiatry Clinic
4. Treatment resistant depression diagnosis confirmed by the ordering physician (treatment failure defined as the lack of clinically meaningful response in depression following an antidepressant trial)
5. Ongoing SI present beyond the screening phase of the study (confirmed with Beck SSI score ≥4).
6. Pass the TMS adult safety screening (TASS) questionnaire
7. Voluntary outpatients capable to consent to treatment and seen at the UC San Diego Health Interventional Psychiatry program.
8. Able to adhere to the treatment schedule.

Exclusion Criteria:

1. Previously undergone the Brief Cognitive Behavioral Therapy for Suicide Prevention (BCBT-SP) protocol
2. Currently undergoing an evidence based psychotherapy treatment (according to the policies by the American Psychological Association)
3. Presence of SI prompting emergent hospital stay (SI in which the participant can maintain voluntary and capable as an outpatient, as well as recent suicide attempt, will not be exclusionary)
4. Not capable to consent to treatment or not suitable for outpatient treatment
5. Have a cardiac pacemaker or implanted medication pump; any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy, cerebral aneurysm, significant head trauma with loss of consciousness for greater than 5 minutes; Have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
6. Based on eligibility for Intranasal Esketamine in the UCSD IPP clinic: Lifetime diagnosis of bipolar I or II disorder or schizophrenia spectrum disorder or current diagnosis of a substance use disorder or cognitive disorder documented in the electronic medical records

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Beck Scale for Suicidal Ideation | 1-week post treatment
TMS-EEG N100 peak | 1-week post treatment

SECONDARY OUTCOMES:
Suicidal Ideation Attributes Scale (SIDAS) | 1-week post treatment
Columbia Suicide Severity Scale (C-SSRS) | 1-week post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Health - 4S Ranch, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided